CLINICAL TRIAL: NCT01882140
Title: The Use of Electrical Stimulation by Capacitive Field in the Repair of Skin Burns and Quality of Life: a Double-blind Randomized Controlled Clinical Trial
Brief Title: The Use of Electrical Stimulation by Capacitive Field in the Repair of Skin Burns and Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, PHD Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1143-4821
Record Dates: First submitted 2013-05-28; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Burns; Wound Healing
Keywords: burns; wound healing; magnetic field therapy
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Experimental): Patients in the Study Group will receive daily treatment for 60 minutes. The treatment is initiated within 24 hours following surgery to achieve graft. Use of Electrical Stimulation by Capacitive Field was the only addition to the current standard of care of the Emergency Unit of HC-FMRP/USP. These Electrical Stimulation by Capacitive Field devices do not produce heat or cause any sensation in tissue. The equipment will produce an electrical stimulation of low intensity pulsed output (1.5 MHz, 1:4 duty cycles, 30mW). The electrodes consist of two metal plates (20x20cm) separated by an insulating material.
  Interventions: Other: Electrical Stimulation by Capacitive Field
- Control Group (Sham devices) (Placebo Comparator): Patients in the control group (Sham group) will receive the same treatment but the device remains off. Use of Electrical Stimulation by Capacitive Field was the only addition to the current standard of care of the Emergency Unit of HC-FMRP/USP.
  Interventions: Other: Electrical Stimulation by Capacitive Field Placebo Sham

INTERVENTIONS:
Other: Electrical Stimulation by Capacitive Field
  Arms: Study Group
Other: Electrical Stimulation by Capacitive Field Placebo Sham
  Arms: Control Group (Sham devices)

SUMMARY:
The high incidence of burn injuries and mortality and morbidity as well as the high economic impact associated with this type of injury justifying the need to develop new technologies for the treatment of burn patients. Electrical stimulation for wound healing is a resource that has been increasingly used in routine physical therapists, but has the disadvantage of needing means of wet contact between the electrode and injury. The other resource used for therapeutic healing is conventional electrical stimulation of low intensity for capacitive field, a technique of physical therapy intervention not commercially available in Brazil. This new technology seems to have significant physiological effects in tissue repair and has been used for the treatment of chronic wounds which healed with difficulty. The objective is to analyze the effects of electrical stimulation of low intensity for capacitive field in healing skin burns. Patients from both genders aged over 18 years who have burns, will be evaluated and treated at the Emergency Unit of the Hospital of the Faculty of Medicine of Ribeirão Preto, University of São Paulo. The stimulation will be initiated within 24 hours after surgery to perform the graft and will be held daily for 60 minutes during the patient's stay or until complete healing of the skin. The electromagnetic field will be placed on the care of the burned area and / or the donor skin graft, not interfering with departmental procedures. Will be performed photographic record standardized wound by a digital camera, and then quantified by a computer program. Expected to reduce the period of hospitalization and thus lowering the cost of treatment, and the possibility of improving the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the Burns Unit of Clinical Hospital, Faculty of Medicine of Ribeirão Preto / USP, in the period between September 2014 and June/2013.
* greater than 18 years.
* deep acute burn requiring excision and grafting

Exclusion Criteria:

* patients who use medicines that may interfere with the process of tissue repair.
* body mass index less than 16 kg / m²
* older than 65 years

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-11 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation of the lesion | Two years
  The following parameters will be documented wound: wound appearance, capillarity, percentage of epithelialization, graft, signs of infection and sensitivity of the wound by burning to touch and clamping.

SECONDARY OUTCOMES:
standard photographs records of the wounds and quantified by ImageJ ® software | Two years
  Will be held the photographic record standardized wound by a digital camera (resolution ≥ 6.0 Megapixel) and subsequently quantified by ImageJ ® software. Each image is calibrated by the tool "Analyze / Set Scale", which allows you to adjust the measure in pixels / cm through the rule contained in the photo. After this standardization selecting the plugin "Polygon" delimiting the border of the lesion with the mouse saving in extension ROI. Then the software automatically calculates the area in cm² (command <CTRL +M>).
quantification of wounds photographs by digital software | Two years
  A computer software CaPAS - Carotid Plaque Analysis Software - will be used for the analysis of two-dimensional images scanned by statistical indexes of the first order (mean gray level and standard deviation) and second order (Entropy, Energy and Homogeneity).

OTHER OUTCOMES:
assessment of health status of burned patients | Two years
  For assessing the health status of burned patients will use a'' Burn Specific Health Scale-Revised'' (BSHS-R) in its version validated for the Portuguese of Brazil.

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Roberto de Jesus Guirro, PHD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.fmrp.usp.br